CLINICAL TRIAL: NCT04565496
Title: An Open Label, Single-arm, Phase 2 Study of Neoadjuvant PEMbrolizumab Before Radical PROstatectomy (PEM-PRO) in High-risk Prostate Cancer Patients
Brief Title: Phase 2 Study of Neoadjuvant PEMbrolizumab Before Radical PROstatectomy in High-risk Prostate Cancer Patients
Acronym: PEM-PRO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Giorgio Gandalgia (Unknown); Alberto Briganti (Unknown); Vito Cucchiara (Unknown)
Responsible Party: Principal Investigator, Francesco Montorsi, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEM-PRO
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab will be administered at the dose of 200 mg intravenously, every 3 weeks, for a total of 3 cycles prior to RP and ePLND
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered at the dose of 200 mg intravenously, every 3 weeks, for a total of 3 cycles prior to RP and ePLND

SUMMARY:
This is a phase 2, open-label, non-randomized, single-arm study in patients with high-risk PCa diagnosed with prostate biopsy and undergoing RP and ePLND. Pembrolizumab will be administered at the dose of 200 mg intravenously, every 3 weeks, for a total of 3 cycles prior to RP and ePLND. Local, nodal and systemic staging with prostate mpMRI, abdominal and chest CT, PSMA-PET/CT and bone scans will be performed before the administration of pembrolizumab. Surgery will be planned at the time of study inclusion to be done within 3 weeks of the last dose of study drug (screening: 3 weeks; cycle 1 followed by 3 weeks; cycle 2 followed by 3 weeks; cycle 3 followed by 3 weeks to surgery = 12 weeks from inclusion to surgery). Patients will receive 3 cycles of pembrolizumab at 200mg 3 weekly prior to RP and ePLND. Surgery will take place within 3 weeks after the last dose of the study drug. After surgery, patients with the evidence of aggressive disease features (namely, pathologic grade group 4-5; pT3b-4 and/or LNI) will be managed according to local guidelines (adjuvant radiotherapy with or without ADT will be allowed). Further Anti PD-1 therapy will not be given post-operatively. PD-L1 status will be retrospectively assessed on both tumour cells and immune cells in tissue specimens from for all patients enrolled in the study.

DETAILED DESCRIPTION:
This is a phase 2, open-label, non-randomized, single-arm study in patients with high-risk PCa diagnosed with prostate biopsy and undergoing RP and ePLND. Screening assessments should be performed no more than 3 weeks prior to the start of study treatment. Local, nodal and systemic staging with prostate mpMRI, abdominal and chest CT, PSMA-PET/CT and bone scans will be performed before the administration of pembrolizumab. Pembrolizumab will be administered at the dose of 200 mg intravenously, every 3 weeks, for a total of 3 cycles prior to RP and ePLND. Following the screening assessment, subsequent assessments will be carried out after the 3 administrations of the study drug prior to RP and ePLND. If an unscheduled assessment is performed and the patient has not progressed, the results should be reported at the next scheduled visit. After the last cycle of pembrolizumab, mpMRI and PSMA-PET/CT scan will be performed to re-stage the tumour. Progressive disease will be defined as an increase of 20% in the maximum diameter of the index lesion at multiparametric MRI or as the onset of nodal or distant metastases at imaging or onset of symptoms and skeletal related events. In the case of symptomatic disease progression (i.e., de novo onset of symptomatic distant metastases), the patient will not complete the 3 cycles of pembrolizumab and will be considered for immediate imaging (i.e., bone scan, mpMRI and PSMA-PET/CT scan) to re-stage the tumour and for treatment according to clinical guidelines. After RP, patients will be managed according to clinical guidelines. PDL-1 status will be assessed on all samples of patients enrolled on the study. Tissue and blood samples will be collected before and after the administration of pembrolizumab. The presence of biomarkers predictive of radiological and pathological response to neoadjuvant administration of pembrolizumab will be assessed. Patients will be monitored carefully for the development of adverse events and will be monitored for clinical evidence of disease progression according to usual standards of clinical practice. Adverse events will be evaluated according to criteria outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. There will be no intrapatient dose escalation in this study. For individual patients that experience dose-limiting toxicities, no criteria for dose modification of pembrolizumab will be applied, but only criteria for dose delays as detailed in the protocol. Patients will be treated with a maximum of 3 cycles of therapy until surgery (i.e. RP and ePLND), provided that no dose-limiting toxicities will occur throughout the treatment course for each individual patient.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of prostate cancer.
2. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
3. PCa detected at prostate biopsy (random biopsy with at least 12 cores taken ± target biopsy according to the mpMRI findings).
4. The participant should be fit and planned for RP and ePLND (according to clinical guidelines).
5. The participant should be affected by high-risk PCa defined as PSA ≥20 ng/ml and/or clinical stage ≥T3 at digital rectal examination and/or biopsy grade group 4-5.
6. No evidence of lymph node invasion (cN0) and metastatic disease (M0) at imaging (mpMRI, PSMA-PET/CT and bone scan).
7. Have provided archival tumour tissue sample or newly obtained core or excisional biopsy of a tumour lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation.
9. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.
10. Willingness to use contraception during study treatment

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
2. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
3. Has received prior surgery or radiotherapy for PCa.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
13. Has a known history of hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
14. Has a known history of active TB (Bacillus Tuberculosis).
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Has a history or current evidence of unstable cardiovascular disease
18. Has a history or current evidence of congestive heart failure
19. Severe hypersensitivity (Grade 3) to pembrolizumab and/or any of its excipients

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients affected by prostate cancer
Enrollment: 59 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node invasion | 12 months
  Reduction by 50% of the rate of lymph node invasion

SECONDARY OUTCOMES:
Pathologic response or presence of minimal residual disease | 12 months
  Absence of morphologically identifiable carcinoma in the prostatectomy specimen or the presence of minimal residual disease (i.e., ≤3 mm maximum diameter of residual tumour in the prostatectomy specimen)
Radiological response | 12 months
  Radiological response will be defined as a tumour reduction of 30% in the maximum diameter of the index lesion as measured by mpMRI
Positive surgical margins | 12 months
  Positive surgical margins at final pathology
PSA persistence or early biochemical recurrence | 36 months
  Postoperative PSA ≥0.1 ng/ml at 6-8 weeks after surgery or two consecutive PSA values ≥0.2 ng/ml within 2 years after surgery
Rate of adverse events | 36 months
  Safety

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No